CLINICAL TRIAL: NCT00279409
Title: Developing More Efficacious Treatments for Children With ADHD Who Are "Partial" or "Non-responders" to Stimulants
Brief Title: Treatment of Children With ADHD Who do Not Fully Respond to Stimulants
Acronym: TREAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment Rate too slow
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Bristol-Myers Squibb (Industry); Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5064; P30MH071478 (NIH)
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Treatment resistant; Partial responder; Non-responder; Atypical Antipsychotic
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Aripiprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aripiprazole (Active Comparator): This treatment arm (also called the "combination arm") consists of parent training plus continued treatment on a stimulant (that is tolerated but has not yet decreased ADHD symptoms enough to meet our criterion of response), plus augmentation with aripiprazole. Aripiprazole pills are taken once daily over a period of 8 weeks, with patients evaluated on a weekly basis. Dosing will start at 2.5 mg and will be titrated up to 5 mg by week 1, and up to 10 mg by week 2 and for the remainder of the trial.
  Interventions: Drug: aripiprazole
- Sugar pill (Placebo Comparator): This treatment arm (also called the "simple treatment" arm) will consist of parent training plus continued treatment on a stimulant (that is tolerated but has not yet decreased ADHD symptoms enough to meet our criterion of response), plus a placebo matching aripiprazole. Placebo pills are taken once daily over a period of 8 weeks, with patients evaluated on a weekly basis.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: aripiprazole — double blind capsules (abilify or placebo) taken once daily, up to 10mg.
  Other Names: Abilify
  Arms: aripiprazole
Drug: Sugar pill — double blind capsules (abilify or placebo) taken once daily, up to 10mg.
  Arms: Sugar pill

SUMMARY:
The purpose of this pilot is to initiate a program of research into the development of effective medication techniques to treat those children with ADHD who are referred because they are "partial" or "non-responders" to standard stimulant treatment.

DETAILED DESCRIPTION:
We propose to do this with a single site, ten week, pilot study of 40 school age children, ages 6-17, with Attention-Deficit/ Hyperactivity Disorder (ADHD) and moderate or greater impairment (C-GAS < 55) who show ADHD symptoms despite a trial in the community with their primary care practitioner with either of two of the most commonly used stimulants (i.e., either OROS-MPH (Concerta) or mixed salts of amphetamine (Adderall-XR)).

These children first will be classified into three groups: Group 1, those who had been treated with a maximal dose of stimulant with partial or no response; Group 2, those treated with a suboptimal dose of stimulant and showing partial or no response, and Group 3, those who developed side effects that limited continued treatment with optimal doses of a stimulant.

The next step will be to enter these children into an open, two week trial to confirm their treatment resistance. Group 2, those treated with suboptimal doses, will have the dosage increased to the maximum recommended stimulant dose. Group 1, those who had been treated for 4 weeks with maximal doses of a stimulant, or Group 3, those who developed moderate to severe drug-related side effects, will be switched to the other class of stimulant for a two week trial, unless they have been tried on both classes. Those children will be maintained on their current class of stimulant for two weeks. At the end of the two weeks, all children will be rated on the ADHD-IV-RS by the Study Doctor. Those who have shown moderate to severe side effects or those who respond will exit the trial and be treated openly. Children from Group 2 who continue to show no improvement after a week will switch to the other stimulant. All children from Group 2 tried on both stimulants and all children from Groups 1 and 3 who continue to show mean scores greater than 1 SD over the mean for age will be referred to Phase 2.

During phase 2, they will be randomized to one of two treatment arms for eight weeks. The first treatment arm, the "simple treatment" arm, will consist of parent training plus continued treatment with a stimulant that is tolerated but has not yet decreased ADHD symptoms enough to meet our criterion of response, plus a placebo matching aripiprazole. The second treatment arm, called the "combination" arm, will consist of parent training plus continued treatment on stimulant plus augmentation with a second generation antipsychotic (aripiprazole). Aripiprazole (Abilify™ ) is a product that is FDA-approved and marketed for the treatment of schizophrenia and for the treatment of acute manic episodes associated with Bipolar I Disorder in adults only. However, aripiprazole is also used to treat children and adolescents with aggressive and oppositional disorders in standard clinical practice. We will continue randomizing patients until we have 40 children with ADHD become eligible to enter Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish speaking parent/guardian. Parent/guardian and child must be able to understand the protocol.
2. Primary diagnosis of ADHD despite treatment with a stimulant by the primary care treatment provider.
3. Non-responder or partial responder to stimulant treatment. ADHD symptoms and clinical impairment despite treatment with stimulant (including OROS-MPH [Concerta] or mixed salts amphetamine [Adderall]).
4. IQ of greater than 70.
5. The subject must be in school.
6. The family must be able to attend weekly visits.

Exclusion Criteria:

1. Unable to understand protocol or follow study procedures.
2. Subject doing well on stimulants.
3. Subjects showing lack of response or minimal response to stimulants due to non-compliance with taking medication or taking suboptimal doses.
4. Autism, Psychosis, Bipolar Disorder, Drug Abuse, significant suicidality, or any other psychiatric disorder (such as MDD, Anxiety Disorders, Eating Disorders) in addition to ADHD that will require treatment with additional medication or therapy.
5. The subject is using or abusing recreational drugs or has a positive urine toxicology screen (except for stimulants).
6. The subject has a history of physical, sexual, or emotional abuse that resulted in a clinically significant impact on clinical presentation, potentially driving some of the symptoms of ADHD.
7. Females who are pregnant or breast-feeding or who have a positive urine pregnancy test.
8. Sexually active females and males who do not agree to use adequate birth control.
9. Abnormal cardiac function.
10. Subject is taking prohibited concomitant medication during phase 1 or phase 2 of the trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence L Greenhill, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole | Sugar Pill
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Despite all efforts to contact the study team members to obtain the data, efforts were unsuccessful. No study data are available
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Sugar Pill | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: ADHD Rating Scale - IV (ADHD-RS-IV)
Time Frame: weekly
Population: as for baseline characteristics
Arm/Group | Aripiprazole | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Despite all efforts to contact the study team members to obtain the data, efforts were unsuccessful. No study data are available
Description: Despite all efforts to contact the study team members to obtain the data, efforts were unsuccessful. No study data are available
Arm/Group | Aripiprazole | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No